CLINICAL TRIAL: NCT02788149
Title: Ultrasound Against Obstructive Sleep Apnea
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Resources did not come to fruition
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Gaurav Chauhan, Resident physician, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: HFHREVIEW
Record Dates: First submitted 2016-05-22; First posted 2016-06-02 (Estimated); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: Ultrasonography; Submental; Lateral Parapharyngeal wall; Tongue base thickness; Polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Ultrasonography; Polysomnography

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STUDY GROUP (Experimental): Model development group: This group will get Ultrasound of neck exam followed by polysomnography. We will use this group to identify the ultrasonographic parameters that have strong association of predicting obstructive sleep apnea. We will use these these predictors to estimate the patient's probability of severe OSA, which then will be used to test the receiver operating characteristic (ROC) curve of diagnosing severe OSA. The optimal cut-off value of the ROC curve will be defined as the one with the least (1 - sensitivity)2+ (1- specificity)2 in the model-development group. This formula will then tested in the validation group.
  Interventions: Device: Ultrasound Exam; Device: Polysomnography
- validation group (Active Comparator): One third patients in the cohort will be randomly assigned to this group. This group will get ultrasound of neck exam followed by polysomnography. The predictors will be tested in his group.
  Interventions: Device: Ultrasound Exam; Device: Polysomnography

INTERVENTIONS:
Device: Ultrasound Exam — Ultrasound of Neck will be used to assess the Lateral parapharyngeal wall thickness. Ultrasound of neck with Submental approach will be used to assess tongue base thickness, subcutaneous fat thickness, retropalatal diameter, retroglossal diameter and upper airway length during normal tidal expiration, forced inspiration and muller's maneuver
  Other Names: Ultrasonography
Device: Polysomnography — Full-night PSG will be performed in the sleep laboratory according to protocol of sleep medicine department after US assessment. Apnea will be defined as the absence of airflow ≥10 sec and hypopnea will be defined as >50% decrease in airflow ≥10 sec associated with reduced arterial oxygen saturation by 4%, or an arousal. These two parameters are collectively defined as apnea-hypopnea index (AHI). An arousal will be recorded if there is a 3-second or longer abrupt shift in electroencephalogram frequency to alpha or theta or above 16 Hz, following at least 10 seconds of sleep, and, if arising in rapid eye movement sleep, there should be a rise in electromyographic tone. An independent technician blinded to the US results will analyze the sleep studies.
  Episodes of AHI per hour will be used to diagnose and grade the severity of OSA:
  Non-OSA : < 5/hr mild OSA : 5- 14/hr moderate OSA :15-29/hr and severe OSA : ≥30/hr.
  Other Names: Sleep Study

SUMMARY:
To investigate the accuracy of neck ultrasound in identifying and discriminating the severity of obstructive sleep apnea (OSA).

Primary objective: To test the hypothesis that ultrasound can be used as a reliable tool for identifying the anatomic characteristics and dynamic changes of pharyngeal airspace in patients with OSA.

Secondary objective: Investigate if ultrasound can be used to discriminate OSA severity.

The investigators will compare these results to the results from polysomnography study.

DETAILED DESCRIPTION:
Investigators are conducting a prospective randomized control trial. Two-thirds of the participants will be randomly selected as the model-development group while the remaining one-third will serve as the validation group. The allocation will be based on a computer-generated random assignment. Ultrasonography and polysomnography operators will be blinded to other results.

Anthropometric Measurements:

Demographic data, including age, gender, weight (kilograms), body height (centimeters) and neck circumference (NC), will be recorded. Weight and height will be recorded with the patients wearing light clothes, but no shoes. Body mass index (BMI) will be then calculated as weight (kg) divided by height squared (mt2). NC will be measured (in cm) with a flexible tape at the level of the cricothyroid membrane after a gentle expiration by the subject while standing upright. History of hypertension, diabetes, hyperlipidemia or any other cardiovascular diseases will be recorded according to medical records or statements by the patients. All participants will be asked to complete the Epworth Sleepiness Scale (ESS), a subjective self-reported measure of excessive daytime sleepiness, within the same session before the ultrasound examination.

Polysomnography :

Full-night polysomnography (PSG) will be performed in the sleep laboratory according to protocol of sleep medicine department after US assessment. Apnea will be defined as the absence of airflow ≥10 sec and hypopnea will be defined as >50% decrease in airflow ≥10 sec associated with reduced arterial oxygen saturation by 4%, or an arousal. These two parameters are collectively defined as apnea-hypopnea index (AHI). An arousal will be recorded if there is a 3 second or longer abrupt shift in electroencephalogram frequency to alpha or theta or above 16 Hertz, following at least 10 seconds of sleep, and, if arising in rapid eye movement sleep, there should be a rise in electromyographic tone. An independent technician blinded to the US results will analyze the sleep studies.

Episodes of AHI per hour will be used to diagnose and grade the severity of OSA:

Non-OSA : < 5/hr mild OSA : 5- 14/hr moderate OSA:15-29/hr and severe OSA : ≥30/hr.

Ultrasonography:

The US will be done by an independent operator. All the measurements will be made by the same operator, who is experienced in US scanning and will be blinded to the polysomnographic data.

Lateral Pharyngeal Wall (LPW) scanning

1. Participants will lay supine on the examination couch. The neck of the participant will be slightly extended, with the infraorbital meatal baseline (the line joining infraorbital margin and ear tragus) perpendicular to the scanning table. A 35° soft pad will be placed under the neck.
2. C5-2 or C7-5 Mega hertz curvilinear transducer will be used. The oblique coronal plane of the parapharyngeal space will be scanned with the transducer longitudinally placed on the lateral side of the neck, just underneath the lateral border of the occipital bone.
3. The long axis of the ipsilateral internal carotid artery will be identified with color application.
4. The distance between the internal carotid artery and the echogenic surface of pharynx will be used to measure the LPW thickness in an oblique coronal plane.
5. All the measurements will be recorded on frozen images when the lateral wall of the pharynx moves farthest away from the transducer (presumably the airway will decrease to its smallest caliber).
6. The maximum thickness of LPW on both sides will be measured 3 times on 3 separate images, and the mean value will be obtained for analysis. Values on both sides of the neck will be summed to determine the total LPW thickness measured by ultrasound.

Submental scanning Before the measurement of dynamic changes, participants will be given time to practice the maneuvers under instruction. Forced inspiration will be desired to approach the inspiratory reserve volume by maximal effort of inspiration within 3 sec. Mullers maneuver (reverse valsalva) will be performed by an attempt at vigorous inhalation with the mouth and nose closed. To localize measurement, two strategies will be applied. First, no shoulder and head movement will be allowed during the maneuver. We will measure the airspace 3 times in every participant based on the same level of US-structure composed of tongue, hypoglossal muscle and geniohyoid muscle and the final recorded value will be mean of the three values.

1. Position and plane of scanning - Investigators will place awake the participant in supine position with infraorbital meatal baseline perpendicular to the scanning table, similar to the position used for lateral pharyngeal wall measurement.
2. Locate the pharynx through HM plane: We will scan from hyoid bone to external auditory meatus (HM plane), at level of oropharynx. The transverse diameter of pharynx will be determined by outer margin of air-column on ultrasound.
3. Measurement of dynamic change of airspace: The probe will be tilted upward and downward gradually to locate Retropalatal (RP) and Retroglossal (RG) in pharynx, defined as air column at the highest plane near the uvula before it was obscured by soft palate & at the plane just above hyoid bone, respectively. The transverse diameters of RP and RG are determined by outer margin of air-column, where they were measured at Muller's maneuver, inspiration and expiration.
4. The midline sagittal plane of the tongue base was scanned with the transducer placed on the submental skin of the neck, between the hyoid bone and the symphysis of the mandible. The operator may tilt the transducer slightly aside to search the hyperechoic raphe of the tongue, which is the landmark of the midline septum of the tongue. The participant will be first instructed to remain still and silent during the measurements and to breathe normally and avoid tongue movement, swallowing or talking. The maximum distance between the submental skin and the dorsal surface of the tongue base, tongue base thickness (TBT eupneic), and subcutaneous fat thickness (SFT - eupneic), were recorded and measured on frozen ultrasound images at the end of expiration during eupneic breathing and during Muller's maneuver.

The TBT and SFT will be recorded and measured on frozen ultrasound images on performance of the MM with the tongue base positioned farthest away from the transducer (i.e. with the pharyngeal airway presumably decreased to its smallest caliber). The maximum TBT and SFT on the Muller's Maneuver (MM) were measured three times on three separate images, and the mean values, TBT (MM) and SFT (MM), will be obtained for analysis. The difference in TBT, TBT (difference), on eupneic breathing and the MM was defined as TBT (MM) - TBT (eupneic). The difference in SFT, SFT (difference), on eupneic breathing and the MM will be defined as SFT (MM) - SFT (eupneic). TBT (difference) and SFT (difference) will be computed for each participant for further analysis.

Reliability Study - To guard against US operator bias fifteen participants will be invited to take part in the reliability study of ultra-sonographic measurement. Participants will be scanned and repositioned by 2 operators independently on the same day for the assessment of inter-operator reliability, and each operator will be blinded to the examination results of the other operator. The participants will be then scanned by the main US operator again 2 to 3 weeks later to determine intra operator reliability. Participants will be provided appropriate fare for their travel.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged ≥18 years-old and who are arranged to receive polysomnography for suspected OSA, as per STOP BANG questionnaire, will be eligible for the study

Exclusion Criteria:

* Refusal to participate
* Inability to perform the maneuvers
* Presence of congestive heart failure
* Presence of chronic pulmonary disease demonstrated on pulmonary function testing
* Active neurologic event
* Active infection or surgery four weeks prior to screening
* Active inflammation in head and neck region
* Burns, trauma, radiotherapy involving head and neck region
* Other diagnosis of sleep disorders
* Ascites, benign or malignant abdominal mass and
* Pregnancy
* Craniofacial abnormalities
* Presence of severe nasal obstruction
* Oral cavity, Oropharyngeal or laryngeal masses
* Cervical rigidity with limited neck flexion and head extension
* No previous diagnosis of OSA or treatment instituted for OSA
* Any patients whose PSG reports had a total sleep time of less than two hours or had no rapid eye movement sleep will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2023-01 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic exam of neck to measure of static and dynamic predictors of obstructive sleep apnea | 1 Year
  Investigators will measure Lateral parapharyngeal wall thickness (cms), upper airway length(cms), tongue base thickness(cms), subcutaneous fat thickness(cms), Retropalatal diameter(cms), Retroglossal diameter(cms) during normal tidal breathing as static indicators. Investigators will also measure tongue base thickness(cms), subcutaneous fat thickness(cms), Retropalatal diameter(cms), Retroglossal diameter (cms) during forced inspiratory maneuver and muller's maneuver as dynamic indicators. All measurements will be taken 3 times and mean will be reported. Investigators will calculate the percentage change in the above mentioned predictors during muller's maneuver Investigator will assess the predictive value of these variables in patients with obstructive sleep apnea, as diagnosed by Polysomnography.
polysomnography | 1 year
  Apnea will be defined as the absence of airflow ≥10 sec and hypopnea will be defined as >50% decrease in airflow ≥10 sec associated with reduced arterial oxygen saturation by 4%, or an arousal. These two parameters are collectively defined as apnea-hypopnea index (AHI).
  Episodes of AHI per hour will be used to diagnose and grade the severity of OSA:
  Non-OSA : < 5/hr, mild OSA : 5- 14/hr, moderate OSA:15-29/hr and severe OSA : ≥30/hr.
Anthropometric measurement | 1 year
  Demographic data, including age, gender, weight (kilograms), body height (centimeters) and neck circumference (NC), will be recorded by a trained assistant in the sleep clinic. Weight and height will be recorded with the patients wearing light clothes, but no shoes. Body mass index (BMI) will be then calculated as weight (kg) divided by height squared (m2). NC will be measured (in cm) with a flexible tape at the level of the cricothyroid membrane after a gentle expiration by the subject while standing upright. History of hypertension, diabetes, hyperlipidemia or any other cardiovascular diseases will be recorded according to medical records or statements by the patients. All participants will be asked to complete the Epworth Sleepiness Scale (ESS), a subjective self-reported measure of excessive daytime sleepiness, within the same session before the ultrasound examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health Systems, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes